CLINICAL TRIAL: NCT06022861
Title: A Randomized, Double-blind, Multicenter, Phase 3 Study to Compare the Efficacy and Safety of LY01015 and Opdivo®（Nivolumab Injection）Combined Respectively With Fluorouracil Plus Cisplatin in Participants With Advanced or Metastatic Esophageal Squamous Cell Carcinoma.
Brief Title: A Study to Compare the Efficacy and Safety of LY01015 and Opdivo® Combined Respectively With Chemotherapy in Advanced or Metastatic Esophageal Squamous Cell Carcinoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shandong Boan Biotechnology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LY01015/CT-CHN-302
Record Dates: First submitted 2023-08-09; First posted 2023-09-05 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Fluorouracil; Cisplatin; Nivolumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LY01015+ Fluorouracil + Cisplatin (Experimental)
  Interventions: Drug: LY01015; Drug: Fluorouracil; Drug: Cisplatin
- Opdivo® + Fluorouracil + Cisplatin (Active Comparator)
  Interventions: Drug: Fluorouracil; Drug: Cisplatin; Drug: Opdivo®

INTERVENTIONS:
Drug: LY01015 — Intravenouslly (IV) 240mg every 2 weeks (Q2W) during the combined chemotherapy period, thereafter, 480mg every 4 weeks(Q4W) during the maintenance treatment period
  Arms: LY01015+ Fluorouracil + Cisplatin
Drug: Fluorouracil — Intravenouslly (IV) l 800mg/m2 every 4 weeks (（on Day 1 through Day 5)during the combined chemotherapy period
Drug: Cisplatin — Intravenouslly (IV) 80mg/m2 every 4 weeks (Q4W) during the combined chemotherapy period
Drug: Opdivo® — Intravenouslly (IV) 240mg every 2 weeks (Q2W) during the combined chemotherapy period, 480mg every 4 weeks(Q4W) during the maintenance treatment period within 24 weeks, thereafter converted to LY01015 480mg every 4 weeks(Q4W).
  Arms: Opdivo® + Fluorouracil + Cisplatin

SUMMARY:
This is a randomized, double-blind, multicenter, Phase 3 study to compare the efficacy and safety of LY01015 and Opdivo®（Nivolumab Injection）combined respectively with fluorouracil plus cisplatin in participants with unresectable advanced, recurrent or metastatic previously untreated esophageal squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to sign the informed consent form.
2. Male or female aged 18 to 75 years patients.
3. Histopathologically confirmed esophagus squamous cell carcinoma.
4. Diagnosed with advanced or metastatic ESCC per AJCC 8th edition, not be amenable to curative approaches( such as definitive chemoradiation/surgery), not received prior systemic anti-cancer therapy for progressive or metastatic disease. Prior neoadjuvant, adjuvant or definitive radiotherapy/chemoradiotherapy/chemotherapy for locally advanced diseases is permitted if time from the last dose to recurrence> 24 weeks.
5. Must have at least one measurable lesion assessed by investigator per RECIST 1.1 criteria .
6. ECOG performance status of 0 to 1.
7. Prior to the first dose, the tumor tissue samples must be provided for PD-L1 expression analysis, and PD-L1 TPS≥1%.
8. Expected survival ≥6 months.
9. Adequate organ function at screening.

Exclusion Criteria:

1. Presence of symptomatic brain metastasis or spinal compression, or history of meningeal metastasis. Patients with asymptomatic brain metastases who have received prior treatment are permitted to enroll if the disease is stable, and corticosteroids have not been required for at least 4 weeks prior to screening. Patients with carcinomatous meningitis are ineligible, regardless of whether the disease is clinically stable or not.
2. With high risks of bleeding or fistula due to apparent tumor invasion to esophagus or adjacent organs.
3. Known endoscopy-confirmed near-complete obstruction requiring interventional therapy or with risk of perforation post stent implantation in the esophagus or trachea.
4. Unstable disease within 6 months prior to signing informed consent form, including but not limited to unstable angina, myocardial infarction, NYHA Class II or higher cardiac failure, severe arrhythmia or cerebrovascular accident (including transient ischemic attacks) requiring treatment, or any other poorly-controlled systemic disease, for example, uncontrolled hypertension (systolic pressure ≥160 mmHg or diastolic pressure≥100 mmHg) despite standard treatment.
5. Received prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137 or anti-CTLA-4 agent or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways.
6. Prior cumulative exposure dose of cisplatin>300 mg/m2 and time from the last dose of cisplatin to randomization ≤12 month.
7. Received a live vaccine within 4 weeks prior to the first dose, or be scheduled to receive a live vaccine during the entire course of the study.
8. Received systemic chemotherapy, targeted therapy, immunosuppressants, immunostimulants, biological agents, Chinese herbal medicines for anti-tumor indications (prescription or medical record required), Chinese patent drug or any other investigational agents or participated in interventional clinical study within 4 weeks (or five half-lives, whichever is longer) prior to the first dose.
9. Other conditions, as determined by the investigator, for example, severe deep vein thrombosis, arterial embolism, hepatic encephalopathy, Child-Pugh grade B or more severe cirrhosis, or other acute or chronic disease, mental illnesses or laboratory abnormalities, which may lead to the following consequences: increase the risks associated with study participation or study drug administration, or interfere with the interpretation of study results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 510 (Estimated)
Dates: Start 2023-10-12 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate(ORR) as assessed by IRC | from baseline to week 16

SECONDARY OUTCOMES:
Objective Response Rate(ORR) as assessed by IRC and investigator | from baseline to week 24
Disease Control Rate (DCR) | up to 2 years
Duration of Response (DOR) | up to 2 years
Progression-Free Survival (PFS) | up to 2 years
16-week Progression-Free Survival Rate | from baseline to week 16
24-week Progression-Free Survival Rate | from baseline to week 16
Overall Survival (OS) | up to 2 years
Incidence and severity of adverse effects (AEs) | up to 2 years
Incidence of Anti-Drug Antibodies (ADA) and Neutralizing Antibodies (Nab) | up to 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, China